CLINICAL TRIAL: NCT02894918
Title: A Randomized, Open-label, Multi-center Clinical Trial to Evaluate Addition of Peginterferon Alfa-2a to CHB Patients Treated With NAs and Achieved HBV DNA<15 IU/ml、HBeAg<100 PEIU/ml、HBsAg Positive and HBsAg<1500 IU/ml.
Brief Title: A Study to Evaluate Addition of Peginterferon Alfa-2a to Chronic Hepatitis B (CHB) Patients Treated With NAs
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Jiashang, M.D., Henan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COMBINE
Record Dates: First submitted 2016-08-31; First posted 2016-09-09 (Estimated); Last update posted 2016-09-12 (Estimated); Status verified 2016-09

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination group (Experimental): Maintain NAs treatment while add 48-week standard treatment by Peginterferon alfa 2a 180µg/week
  Interventions: Drug: Peginterferon alfa-2a
- Mono NA group (No Intervention): Maintain NAs mono-therapy oral-daily for 48 weeks.

INTERVENTIONS:
Drug: Peginterferon alfa-2a — 180ug/0.5ml,hypodermic injection once a week
  Other Names: Pegasys
  Arms: Combination group

SUMMARY:
This study evaluates whether addition of Peginterferon alfa-2a to CHB Patients Treated with nucleoside analogues (NAs) can enhance the rate of HBsAg clearance at end of treatment. This study is a Randomized, open-label, multi-center study.

The CHB patients with NAs treatment and have achieved HBV DNA <15 IU/ml、HBeAg <100 PEIU/ml、HBsAg positive and HBsAg<1500 IU/ml will be randomized into 2 groups:

Group 1 (Combination group): Maintain NAs treatment while add 48-week standard treatment by Peginterferon alfa 2a 180µg/week Group 2 (Mono NA group) : Maintain NAs treatment for 49 weeks. Note: NAs including: LAM, ADV, ETV, or TDF.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients >18 and ≤65 years of age;
* Diagnosed chronic hepatitis B (HBsAg(+) for over 6 months before nucleos(t)ide analogues treatment)
* Patients had achieved HBV DNA<15 IU/ml、HBeAg<100 PEIU/ml、HBsAg positive and HBsAg<1500 IU/ml on treatment of Nucleoside (acid) Analogues (including LAM, ADV, ETV, and TDF )

Exclusion Criteria:

* Decompensated liver disease: including ascites, hepatic encephalopathy, esophagogastric-varicosis and fissure bleeding and other decompensated complication;
* Hypersensitive to interferon(IFN) or its active substance, and ineligible to IFN;
* A history of immunoregulation drug therapy within 1 year before entry including IFN and so on;
* Coinfection with HAV、HCV、HDV、HEV 、HIV or with Other chronic liver diseases such as Alcoholic Liver Disease,Inherited Metabolic Liver Disease,Drug induced Liver Disease and nonalcoholic fatty liver, autoimmune disease including autoimmune hepatitis and Psoriasis and so on;
* Hepatocellular carcinoma(HCC) or alpha feto protein(AFP) levels more than 100ng/ml and Hepatic malignant potential of Imaging examination or AFP levels more than 100 ng/ml for 3 months;
* A neutrophil count of less than 1500 per cubic millimeter or a platelet count of less than 90,000 per cubic millimeter;
* A serum creatinine level that was more than 1.5 times the upper limit of the normal range;
* With other malignant tumors(exclude the cured ones);
* Severe organ dysfunction;
* With severe psychiatric condition or nervous disease such as epilepsy, depression, mania, epilepsy, schizophrenia and so on;
* Uncontrolled diabetes, hypertension or thyroid disease;
* Pregnant women and lactating women or patients with pregnancy plans and not willing to use contraception during the study period;
* Participate in other clinical studies at the same time;
* Patients unsuitable for the research;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-06 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
The rate of HBsAg loss | 48 weeks
  To determine the response rate will be evaluated by HBsAg loss defined as HBsAg level lower than 0.05 IU/ml after 48 week treatment, compared with control group.

SECONDARY OUTCOMES:
Decline of HBeAg quantification | 12 weeks, 24 weeks, 48 weeks of treatment
  Quantitative HBeAg reduction at Weeks 12, 24 and 48 compared with baseline level. Quantitative HBeAg value unit was calculated using 'Paul Ehrlich Institute units per millilitre' (PEIU/ml).
Decline of HBsAg quantification | 12 weeks, 24 weeks, 48 weeks of treatment
  Quantitative HBsAg reduction at Weeks 12, 24 and 48 compared with baseline level. Quantitative HBsAg calculated using 'International Units Per Millilitre' (IU/mL).
The rate of HBeAg loss | 48 weeks
The rate of HBeAg seroconversion | 48 weeks
The rate of HBsAg seroconversion | 48 weeks
Sustained virological response rate | 12 weeks, 24 weeks, 48 weeks of treatment
  Sustained virological response rate will be presented as rate of HBV DNA <15 IU/ml

CONTACTS AND LOCATIONS:
Overall Officials: Jia Shang, M.D., Principal Investigator — Henan People's hospital
Locations (5):
- China (5):
  - Kaifeng Central Hospitl, Kaifeng, Henan
  - Weishi County People's Hospital, Kaifeng, Henan
  - Luoyang Central Hospital, Luoyang, Henan
  - Shangqiu No.1 People's Hospital, Shangqiu, Henan
  - Henan People's Hospital, Zhengzhou, Henan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ott JJ, Stevens GA, Groeger J, Wiersma ST. Global epidemiology of hepatitis B virus infection: new estimates of age-specific HBsAg seroprevalence and endemicity. Vaccine. 2012 Mar 9;30(12):2212-9. doi: 10.1016/j.vaccine.2011.12.116. Epub 2012 Jan 24. PMID 22273662
- [Result] Lu FM, Zhuang H. Management of hepatitis B in China. Chin Med J (Engl). 2009 Jan 5;122(1):3-4. No abstract available. PMID 19187608
- [Result] European Association For The Study Of The Liver. EASL clinical practice guidelines: Management of chronic hepatitis B virus infection. J Hepatol. 2012 Jul;57(1):167-85. doi: 10.1016/j.jhep.2012.02.010. Epub 2012 Mar 20. No abstract available. PMID 22436845
- [Result] Lai CL, Gane E, Liaw YF, Hsu CW, Thongsawat S, Wang Y, Chen Y, Heathcote EJ, Rasenack J, Bzowej N, Naoumov NV, Di Bisceglie AM, Zeuzem S, Moon YM, Goodman Z, Chao G, Constance BF, Brown NA; Globe Study Group. Telbivudine versus lamivudine in patients with chronic hepatitis B. N Engl J Med. 2007 Dec 20;357(25):2576-88. doi: 10.1056/NEJMoa066422. PMID 18094378
- [Result] Liaw YF, Gane E, Leung N, Zeuzem S, Wang Y, Lai CL, Heathcote EJ, Manns M, Bzowej N, Niu J, Han SH, Hwang SG, Cakaloglu Y, Tong MJ, Papatheodoridis G, Chen Y, Brown NA, Albanis E, Galil K, Naoumov NV; GLOBE Study Group. 2-Year GLOBE trial results: telbivudine Is superior to lamivudine in patients with chronic hepatitis B. Gastroenterology. 2009 Feb;136(2):486-95. doi: 10.1053/j.gastro.2008.10.026. Epub 2008 Nov 1. PMID 19027013
- [Result] Marcellin P, Heathcote EJ, Buti M, Gane E, de Man RA, Krastev Z, Germanidis G, Lee SS, Flisiak R, Kaita K, Manns M, Kotzev I, Tchernev K, Buggisch P, Weilert F, Kurdas OO, Shiffman ML, Trinh H, Washington MK, Sorbel J, Anderson J, Snow-Lampart A, Mondou E, Quinn J, Rousseau F. Tenofovir disoproxil fumarate versus adefovir dipivoxil for chronic hepatitis B. N Engl J Med. 2008 Dec 4;359(23):2442-55. doi: 10.1056/NEJMoa0802878. PMID 19052126
- [Result] Chang TT, Gish RG, de Man R, Gadano A, Sollano J, Chao YC, Lok AS, Han KH, Goodman Z, Zhu J, Cross A, DeHertogh D, Wilber R, Colonno R, Apelian D; BEHoLD AI463022 Study Group. A comparison of entecavir and lamivudine for HBeAg-positive chronic hepatitis B. N Engl J Med. 2006 Mar 9;354(10):1001-10. doi: 10.1056/NEJMoa051285. PMID 16525137
- [Result] Moucari R, Korevaar A, Lada O, Martinot-Peignoux M, Boyer N, Mackiewicz V, Dauvergne A, Cardoso AC, Asselah T, Nicolas-Chanoine MH, Vidaud M, Valla D, Bedossa P, Marcellin P. High rates of HBsAg seroconversion in HBeAg-positive chronic hepatitis B patients responding to interferon: a long-term follow-up study. J Hepatol. 2009 Jun;50(6):1084-92. doi: 10.1016/j.jhep.2009.01.016. Epub 2009 Mar 9. PMID 19376603
- [Result] Marcellin P, Bonino F, Yurdaydin C, Hadziyannis S, Moucari R, Kapprell HP, Rothe V, Popescu M, Brunetto MR. Hepatitis B surface antigen levels: association with 5-year response to peginterferon alfa-2a in hepatitis B e-antigen-negative patients. Hepatol Int. 2013 Mar;7(1):88-97. doi: 10.1007/s12072-012-9343-x. Epub 2012 Mar 23. PMID 23518903
- [Result] Chevaliez S, Hezode C, Bahrami S, Grare M, Pawlotsky JM. Long-term hepatitis B surface antigen (HBsAg) kinetics during nucleoside/nucleotide analogue therapy: finite treatment duration unlikely. J Hepatol. 2013 Apr;58(4):676-83. doi: 10.1016/j.jhep.2012.11.039. Epub 2012 Dec 3. PMID 23219442
- [Result] Micco L, Peppa D, Loggi E, Schurich A, Jefferson L, Cursaro C, Panno AM, Bernardi M, Brander C, Bihl F, Andreone P, Maini MK. Differential boosting of innate and adaptive antiviral responses during pegylated-interferon-alpha therapy of chronic hepatitis B. J Hepatol. 2013 Feb;58(2):225-33. doi: 10.1016/j.jhep.2012.09.029. Epub 2012 Oct 6. PMID 23046671
- [Result] Chen J, Wang Y, Wu XJ, Li J, Hou FQ, Wang GQ. Pegylated interferon alpha-2b up-regulates specific CD8+ T cells in patients with chronic hepatitis B. World J Gastroenterol. 2010 Dec 28;16(48):6145-50. doi: 10.3748/wjg.v16.i48.6145. PMID 21182232
- [Result] Lau GK, Piratvisuth T, Luo KX, Marcellin P, Thongsawat S, Cooksley G, Gane E, Fried MW, Chow WC, Paik SW, Chang WY, Berg T, Flisiak R, McCloud P, Pluck N; Peginterferon Alfa-2a HBeAg-Positive Chronic Hepatitis B Study Group. Peginterferon Alfa-2a, lamivudine, and the combination for HBeAg-positive chronic hepatitis B. N Engl J Med. 2005 Jun 30;352(26):2682-95. doi: 10.1056/NEJMoa043470. PMID 15987917
- [Result] Liaw YF, Jia JD, Chan HL, Han KH, Tanwandee T, Chuang WL, Tan DM, Chen XY, Gane E, Piratvisuth T, Chen L, Xie Q, Sung JJ, Wat C, Bernaards C, Cui Y, Marcellin P. Shorter durations and lower doses of peginterferon alfa-2a are associated with inferior hepatitis B e antigen seroconversion rates in hepatitis B virus genotypes B or C. Hepatology. 2011 Nov;54(5):1591-9. doi: 10.1002/hep.24555. PMID 22045673
- [Result] Ning Q, Han M, Sun Y, Jiang J, Tan D, Hou J, Tang H, Sheng J, Zhao M. Switching from entecavir to PegIFN alfa-2a in patients with HBeAg-positive chronic hepatitis B: a randomised open-label trial (OSST trial). J Hepatol. 2014 Oct;61(4):777-84. doi: 10.1016/j.jhep.2014.05.044. Epub 2014 Jun 7. PMID 24915612
- [Result] Ren H, Hu P, Jia S. et al. A multi-center randomized study on the efficacy and safety of switching to peginterferon a-2a(40KD) for 48 or 96 weeks in HBeAg positive CHB patients with a prior NUC history for 1-3 years: an interim analysis of NEW SWITCH study. 2014 AASLD. LB10.
- [Result] 李国军，喻一奇，等。乙型肝炎表面抗原水平对核苷(酸)类似物序贯联合聚乙二醇干扰素a-2a治疗慢性乙型肝炎患者的疗效预测。中华传染病杂志2014.32（2）:100-106
- [Result] Chi H, Xie Q, Zhang NP. et al. Addition of Peginterferon Alfa-2b During Long-term Nucleos(t)ide Analogue Therapy Increases HBeAg Seroconversion and HBsAg Decline - Week 48 Results From a Multicenter Randomized Controlled Trial (PEGON Study). 2014 AASLD ab.1882.
- [Result] Marc Bourlière, Pascaline Rabiega. et al. HBsAg clearance after addition of 48 weeks of PEGIFN in HBeAg negative CHB patients on Nucleos(t)ide therapy with undetectable HBV DNA for at least one year: a multicenter randomized controlled phase III trial ANRS-HB06 PEGAN study: preliminary findings. 2014 AASLD ab1863.
- [Result] Lozano R, Naghavi M, Foreman K, Lim S, Shibuya K, Aboyans V, Abraham J, Adair T, Aggarwal R, Ahn SY, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Barker-Collo S, Bartels DH, Bell ML, Benjamin EJ, Bennett D, Bhalla K, Bikbov B, Bin Abdulhak A, Birbeck G, Blyth F, Bolliger I, Boufous S, Bucello C, Burch M, Burney P, Carapetis J, Chen H, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahodwala N, De Leo D, Degenhardt L, Delossantos A, Denenberg J, Des Jarlais DC, Dharmaratne SD, Dorsey ER, Driscoll T, Duber H, Ebel B, Erwin PJ, Espindola P, Ezzati M, Feigin V, Flaxman AD, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabriel SE, Gakidou E, Gaspari F, Gillum RF, Gonzalez-Medina D, Halasa YA, Haring D, Harrison JE, Havmoeller R, Hay RJ, Hoen B, Hotez PJ, Hoy D, Jacobsen KH, James SL, Jasrasaria R, Jayaraman S, Johns N, Karthikeyan G, Kassebaum N, Keren A, Khoo JP, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lipnick M, Lipshultz SE, Ohno SL, Mabweijano J, MacIntyre MF, Mallinger L, March L, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGrath J, Mensah GA, Merriman TR, Michaud C, Miller M, Miller TR, Mock C, Mocumbi AO, Mokdad AA, Moran A, Mulholland K, Nair MN, Naldi L, Narayan KM, Nasseri K, Norman P, O'Donnell M, Omer SB, Ortblad K, Osborne R, Ozgediz D, Pahari B, Pandian JD, Rivero AP, Padilla RP, Perez-Ruiz F, Perico N, Phillips D, Pierce K, Pope CA 3rd, Porrini E, Pourmalek F, Raju M, Ranganathan D, Rehm JT, Rein DB, Remuzzi G, Rivara FP, Roberts T, De Leon FR, Rosenfeld LC, Rushton L, Sacco RL, Salomon JA, Sampson U, Sanman E, Schwebel DC, Segui-Gomez M, Shepard DS, Singh D, Singleton J, Sliwa K, Smith E, Steer A, Taylor JA, Thomas B, Tleyjeh IM, Towbin JA, Truelsen T, Undurraga EA, Venketasubramanian N, Vijayakumar L, Vos T, Wagner GR, Wang M, Wang W, Watt K, Weinstock MA, Weintraub R, Wilkinson JD, Woolf AD, Wulf S, Yeh PH, Yip P, Zabetian A, Zheng ZJ, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Global and regional mortality from 235 causes of death for 20 age groups in 1990 and 2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2095-128. doi: 10.1016/S0140-6736(12)61728-0. PMID 23245604